CLINICAL TRIAL: NCT01323465
Title: A Phase I, Open-label, Randomised, Crossover Study in 3 Parallel Groups to Evaluate the Effect of Rifampicin, Ketoconazole, and Omeprazole on the Pharmacokinetics of Sativex in Healthy Volunteers
Brief Title: Study to Evaluate the Effect of Rifampicin, Ketoconazole, and Omeprazole on the Pharmacokinetics of Sativex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GWCP0602
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Evaluation of Pharmacokinetics of Sativex in the Absence and Presence of a Known Inducer of CYP3A4; Evaluation of Pharmacokinetics of Sativex in the Absence and Presence of a Potent Inhibitor of CYP3A4; Evaluation of Pharmacokinetics of Sativex in the Absence and Presence of a CYP2C19 Inhibitor
Keywords: Sativex; Cytochrome P450; Pharmacokinetics; Cannabinoids; ketoconazole; omeprazole; rifampicin
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Rifampin; Ketoconazole; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1A (Experimental): Sativex and rifampicin
  Interventions: Drug: Sativex and rifampicin
- Sequence 1B (Experimental): Sativex and rifampicin
  Interventions: Drug: Sativex and rifampicin
- Sequence 2C (Experimental): Sativex and ketoconazole
  Interventions: Drug: Sativex and ketoconazole
- Sequence 2D (Experimental): Sativex and ketoconazole
  Interventions: Drug: Sativex and ketoconazole
- Sequence 3E (Experimental): Sativex and omeprazole
  Interventions: Drug: Sativex and omeprazole
- Sequence 3F (Experimental): Sativex and omeprazole
  Interventions: Drug: Sativex and omeprazole

INTERVENTIONS:
Drug: Sativex and rifampicin — Single dose of 4 sprays Sativex on Day 1, Rifampicin 2 x 300 mg capsules on Days 2-10, Sativex dose of 4 sprays and rifampicin 2 x 300 mg capsules on Day 11.
  Arms: Sequence 1A
Drug: Sativex and rifampicin — Rifampicin 2 x 300 mg capsules on Days 1-9, Sativex x 4 sprays and rifampicin 2 x 300 mg capsules on Day 10, Single dose of Sativex 4 sprays on Day 18.
  Arms: Sequence 1B
Drug: Sativex and ketoconazole — Single dose of 4 sprays Sativex on Day 1, ketoconazole 2 x 200 mg tablets on Days 2-5, Sativex x 4 sprays and ketoconazole 2 x 200mg on Day 6.
  Arms: Sequence 2C
Drug: Sativex and ketoconazole — Ketoconazole 2 x 200 mg tablets on Days 1-4, Sativex x 4 sprays and ketoconazole 2 x 200 mg tablets on Day 5, Single dose of 4 sprays Sativex on Day 9.
  Arms: Sequence 2D
Drug: Sativex and omeprazole — Single dose of 4 sprays of Sativex on Day 1 Omeprazole 2 x 20 mg on Days 2-6. Sativex x 4 sprays and omeprazole 2 x 20 mg on Day 9.
  Arms: Sequence 3E
Drug: Sativex and omeprazole — Omeprazole 2 x 20 mg on Days 1-5, Sativex x 4 sprays and omeprazole 2 x 20 mg on Day 6, Single dose of 4 sprays Sativex on Day 9.
  Arms: Sequence 3F

SUMMARY:
Study to assess the effect of rifampicin, ketoconazole and omeprazole on the pharmacokinetics of a single dose of Sativex and to evaluate the safety of Sativex when given in combination with these other drugs.

DETAILED DESCRIPTION:
An open-label, randomised, crossover, drug interaction study. Subjects were divided into three groups and within each group, subjects were randomised to one of two treatment sequences. Subjects received 4 sprays of Sativex alongside either doses of rifampicin, ketoconazole or omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 45 years of age (inclusive).
* Subjects body mass index was between 18-30 kg/m2 (inclusive) as calculated by: Weight (kg)/height (m2).
* No clinically significant abnormal findings on the physical examination, ECG, medical history, or clinical laboratory results during screening.
* Subjects were to, in the opinion of the investigator, have no clinically significant abnormal findings of renal and hepatic function as determined by serum creatinine, total bilirubin, and transaminase levels.
* Subjects were to be non-users of tobacco products (minimum of 6 months prior to the start of the study).
* Subjects were to have a negative screen for HIV I and II, HBsAg. and antibody to hepatitis C.
* Subjects were to have a negative urine screen for alcohol, drugs of abuse (screening only), and cotinine.
* Subjects were to use an appropriate barrier method of contraception (condom and spermicide) in addition to having their female partner use another form of barrier contraception (e.g. female condom or occlusive cap [diaphragm or cervical vault/caps] with spermicide) during the study and for 3 months following administration of the study drug.
* Subjects were to be able to comply with the protocol and the restrictions and the assessments therein.
* Subjects were to give voluntary written informed consent to participate in the trial.

Exclusion Criteria:

* Subjects were not to have a history or presence of significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* Subjects were not to have any history or presence of family history of schizophrenia, other psychotic illness, severe personality disorder, depression, or other significant psychiatric disorder.
* Subjects were not to have a postural drop of 20 mmHG or more in systolic blood pressure at screening.
* Subjects were not to have participated in a previous clinical trial within 90 days prior to study initiation.
* Subjects were not to have donated plasma within 90 days prior to study initiation.
* Subjects were not to have donated blood within 90 days prior to study initiation.
* Subjects were not to have had an abnormal diet or substantial changes in eating habits within 30 days prior to study initiation.
* Subjects were not to have had treatment with any known enzyme-altering agents (barbiturates, phenothiazines, cimetidine etc.) within 30 days prior to or during the study.
* Subjects were to have no history of known hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
* Subjects were not to use any prescription medication within 14 days prior to or during the study.
* Subjects were not to use any over-the-counter medication within 7 days prior to or during the study.
* Subjects were not to have a history of alcohol or drug abuse within 2 years prior to the study (subjects with a history of previous use of cannabis were not excluded unless they had used cannabis or cannabinoid based medicine within 30 days prior to study drug administration or were unwilling to abstain for the duration of the study).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic analysis - Cmax of Sativex® alone and of Sativex® with concomitant administration of rifampicin, ketoconazole, and omeprazole | Up to Day 8
Pharmacokinetic analysis - AUC(0-t) of Sativex® alone and of Sativex® with concomitant administration of rifampicin, ketoconazole, and omeprazole | Up to day 8
Pharmacokinetic analysis - AUC(0-inf) of Sativex® alone and of Sativex® with concomitant administration of rifampicin, ketoconazole, and omeprazole | Up to Day 8

SECONDARY OUTCOMES:
Adverse Events | Up to follow up, Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit, Quintiles Ltd., London, United Kingdom

REFERENCES:
- [Result] Stott C, White L, Wright S, Wilbraham D, Guy G. A Phase I, open-label, randomized, crossover study in three parallel groups to evaluate the effect of Rifampicin, Ketoconazole, and Omeprazole on the pharmacokinetics of THC/CBD oromucosal spray in healthy volunteers. Springerplus. 2013 May 24;2(1):236. doi: 10.1186/2193-1801-2-236. Print 2013 Dec. PMID 23750331